CLINICAL TRIAL: NCT01525043
Title: Randomized, Parallel-Group, Open Label, Dose Finding Study to Evaluate the Efficacy of Synera Patch Compared to Naproxen Sodium for the Treatment of Lateral and Medial Epicondylitis of the Elbow
Brief Title: Study to Evaluate the Efficacy of the Synera Patch Compared to Naproxen Sodium for Epicondylitis of the Elbow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYN-EPI-2011
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Epicondylitis of the Elbow
Keywords: Epicondylitis
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- Synera single patch applied for 12 hrs/day (Experimental)
  Interventions: Drug: Synera patch for 12hrs/day; Drug: Synera
- Synera sinlgle patch applied for 4hrs twice daily (Experimental)
  Interventions: Drug: Synera patch twice daily; Drug: Synera

INTERVENTIONS:
Drug: Naproxen — Naproxen 500mg BID for the first 2 weeks
  Arms: Naproxen
Drug: Synera patch twice daily — 1 synera patch to cover the treatment area applied for 4 hours, twice daily for the first 2 weeks
  Arms: Synera sinlgle patch applied for 4hrs twice daily
Drug: Synera patch for 12hrs/day — 1 synera patch to cover the treatment area applied for 12 hours, daily for the first 2 weeks
  Arms: Synera single patch applied for 12 hrs/day
Drug: Naproxen — 500mg bid
  Arms: Naproxen
Drug: Synera — Topical appication of single patch to elbow for 12hrs/day
  Arms: Synera single patch applied for 12 hrs/day
Drug: Synera — Single patch applied to elbow for 4hrs/twice daily
  Arms: Synera sinlgle patch applied for 4hrs twice daily

SUMMARY:
The purpose of the this study is to evaluate the sfaety and efficacy of Synera(R)for patients with lateral and medial epicondylitis and compare it to Naproxen sodius.

DETAILED DESCRIPTION:
The objective of this single center is to evaluate the safety and efficacy of Synera ® in lateral and medial epicondylitis . This is an open-label, comaparative study study where the subjects will be randomized to one of the following groups:

1. Synera patch ®: A single patch applied for 4 hours twice daily approximatey 12 hrs apart to the medial or lateral side of the index elbow
2. Synera patch ®: A single patch applied for 12 hours/day to the medial or lateral side of the index elbow
3. Naproxen Sodium: 500mg bid

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical evidence of lateral or medial epicondylitis of the elbow.
* Age 18 or higher
* Minimum of 4 on Question 5 of BPI

Exclusion Criteria:

* Peripheral neuropathy of any origin in the index limb
* Cubital tunnel syndrome in patients with medial epicondylitis
* Cortisone injection in the last 4 weeks into the index limb
* Surgical intervention in the past for the epicondiitis
* Participants in any other clinical trial in the last 30 days
* Known allergy to lidocaine, tetracaine, NSAIDs or PABA
* Uncontrolled pain in the upper extremity or neck that may interfere with evaluation of study drug's response as deemed by the investigator
* Patient who is deemed to be medically unstable by the principal investigator including but not limited to Liver disease or Cardiac arrhythmias
* Patients who are pregnant, lactating or breast feeding
* Vaccination within the last weeks or planning on any vaccinations during the study or for 4 weeks after the study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline recorded at 2 week visit for the question #5 of Brief Pain Inventory (BPI )Scale ® recorded before going to sleep daily | Day 1 and Day 14
  Brief Pain Inventory (BPI )Scale ® recorded before going to sleep daily by the subject and the answer for question 5 is the basis for primary end poit

SECONDARY OUTCOMES:
Pain quality assessment scale | Every visit from the entry
  It is a vlaidated measure to assess the qulaity of scale

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research Institute, Inc.
Locations (1):
- International Clinical Research Institute, Overland Park, Kansas, United States